CLINICAL TRIAL: NCT00002248
Title: A Randomized, Multicenter, Double-Blind, Parallel-Group, Placebo-Controlled Trial of the Efficacy and Safety of Bovine Anti-Cryptosporidium Immunoglobulin (BACI) in the Treatment of Cryptosporidium Enteritis in AIDS Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Univax Biologics Inc (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 081A; UNX-4101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-04

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Antidiarrheals; Cryptosporidiosis; Diarrhea; Acquired Immunodeficiency Syndrome; Cryptosporidium; Immunization, Passive
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; Diarrhea; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: Cryptosporidium Immune Whey Protein Concentrate (Bovine)

SUMMARY:
PRIMARY: To assess the effect of bovine anti-Cryptosporidium immunoglobulin (BACI) on the volume of diarrhea due to Cryptosporidium parvum in AIDS patients who have protracted Cryptosporidium enteritis.

SECONDARY: To assess changes in stool consistency and frequency, body weight, and safety in this patient population.

DETAILED DESCRIPTION:
Forty patients are randomized to receive either BACI or placebo (bovine colostrum from non-immunized cattle) for 1 week. The double-blind portion of the study will be followed by an open-label phase in which all 40 patients receive BACI for 1 week.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antidiarrheal compounds (if dose remains stable).
* Zidovudine (AZT), dideoxyinosine (ddI), dideoxycytidine (ddC), or alternative HIV therapy (provided dose was stable for at least 4 weeks prior to study entry).

Patients must have:

* AIDS.
* Cryptosporidium parvum enteritis.
* Chronic diarrhea.
* Life expectancy of at least 4 weeks.
* Ability to tolerate food by mouth.
* Ability to take the histamine H2-receptor antagonist famotidine (Pepcid).

Prior Medication:

Allowed:

* Antidiarrheal compounds (provided dose has remained stable in the 7 days prior to study entry).
* Zidovudine (AZT), dideoxyinosine (ddI), dideoxycytidine (ddC), or alternative HIV therapy (provided dose has remained stable for at least 4 weeks prior to study entry).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Concurrent unresolved clinical infections with enteric pathogens other than C. parvum (e.g., rotavirus, Salmonella, Shigella, Campylobacter, Giardia, C. difficile toxin, Yersinia, amebiasis, MAI, CMV, Microsporida) as determined by history or routine microbiology screening.
* Other acute infections or concurrent immediately life-threatening medical crisis other than cryptosporidiosis.
* Grossly bloody diarrhea.
* Known allergy to milk or milk products (other than lactose intolerance).

Prior Medication:

Excluded:

* Other experimental therapy (e.g., macrolide antibiotics, paromomycin) within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Gabin Med Group, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - New England Med Ctr, Boston, Massachusetts
  - Saint Elizabeth's Hosp, Boston, Massachusetts
  - Cornell Univ Med Ctr, New York, New York

REFERENCES:
- [Background] Nord J, Ma P, Tacket CO, Dijohn D, Tzipori S, Sahner D, Shieb G. Treatment of AIDS associated cryptosporidiosis with hyperimmune colostrum from cows vaccinated with cryptosporidium. Int Conf AIDS. 1989 Jun 4-9;5:656 (abstract no C586)